CLINICAL TRIAL: NCT02955485
Title: A Prediction Model for Chronic Ankle Instability: Indications for Early Surgical Treatment? An Observational Prospective Cohort
Brief Title: A Prediction Model for Chronic Ankle Instability
Acronym: Predict
Status: Terminated | Type: Observational
Why Stopped: Inclusion issues, not able to include sufficient patients
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Slotervaart Hospital (Other); Amsterdam UMC, location VUmc (Other); Flevoziekenhuis (Other)
Responsible Party: Principal Investigator, Gwendolyn Vuurberg, Gwendolyn Vuurberg, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: W16_258#16.303
Record Dates: First submitted 2016-11-01; First posted 2016-11-04 (Estimated); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Chronic Ankle Instability
Keywords: Ankle; Instability; Prediction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with chronic ankle instability: All patients that develop chronic ankle instability after an ankle sprain and reporting at the emergency department. Experiencing persisting complaints of instability for more than 6 months.
  Interventions: Other: Patients do not undergo any type of interventions, but standard care if offered and accepted.
- Patients without chronic ankle instability: All patients that do not develop chronic ankle instability after an ankle sprain and reporting at the emergency department. Complaints resolve within 6 months.
  Interventions: Other: Patients do not undergo any type of interventions, but standard care if offered and accepted.

INTERVENTIONS:
Other: Patients do not undergo any type of interventions, but standard care if offered and accepted.

SUMMARY:
Chronic ankle instability is a common problem that may follow an ankle sprain. Until a patient has developed chronic ankle instability they are ineligible for surgical treatment although early surgical treatment yields better results compared to surgical treatment of subjects that have experienced recurrent ankle sprains. However, treating all patients with an ankle sprain surgically is not an option due to the high amount of unnecessary invasive interventions.

The objective of this study is to identify which patients will develop chronic ankle instability and to develop a model to predict which patients should receive early surgical treatment.

In this prospective observational cohort all patients (older than 18 years) that report at the emergency department of the participating hospitals after a lateral ankle sprain, of whom an x-ray is made after positive Ottawa Ankle Rules and on which there is no visible fracture or other pathology.

The main study parameter is a significant difference in patient characteristics, foot and ankle configuration and joint pathology between patients who develop chronic ankle instability and patients who do not experience recurrent ankle sprains and restriction during daily live after an initial sprain.

ELIGIBILITY:
Inclusion Criteria:

* At least 16 years old
* Visited the ER within one week after a lateral ankle sprain
* An anteroposterior and lateral x-ray have been made
* Agreed with being approached for this study
* Questionnaires have been returned within 4 weeks
* Reported lateral ankle pain after an ankle sprain or ankle distortion ankle

Exclusion Criteria:

* Present fracture or other joint pathology/bone matrix pathology
* A diagnosed osteochondral defect after primary inclusion
* Medial ankle instability
* Previous ankle surgery
* An unreliable x-ray due to the angle in which it is made or low quality
* Acute surgical repair of the anterior talofibular ligament and/or calcaneofibular ligament or another form of surgery within 6 months after the initial ankle sprain

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients reporting at the ED in the AMC after an ankle sprain are eligible for inclusion. Their condition may vary from a severe sprain to an ankle fracture. All patients will be checked for ankle fractures using the Ottawa Ankle Rules (OAR). In 5-20% of cases a fracture is present with positive OAR, or there is doubt on the presence of a fracture and an x-ray will be taken. However there is always a chance of false positive results on the OAR. In these cases there is may have been a severe ankle sprain without intraarticular pathology visible on the x-ray. These are concluded to be severe sprain cases the investigators will extract for this study to include them in a questionnaire follow-up on the development of CAI.
Sampling Method: Probability Sample
Enrollment: 460 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is a prediction model based several factors. One of these is ankle joint alignment. | 2 years anticipated
  Ankle alignment is assessed as the medial distal tibial angle on a standard anteroposterior x-ray
The primary outcome measure is a prediction model based several factors. One of these is fibular position in relation to the tibia. | 2 years anticipated
  Position of the fibula is assessed on a lateral x-ray.
The primary outcome measure is a prediction model based several factors. One of these is the tibiotalar contact ratio. | 2 years anticipated
  The tibiotalar contact ratio is assessed as an angle originating from the center of the talus to the anterior and posterior edges of the distal tibia.
The primary outcome measure is a prediction model based several factors. One of these is sex. | 2 years anticipated
  Sex is registrated as male-female and has proven to be of prognostic value in previous research
The primary outcome measure is a prediction model based several factors. One of these is height. | 2 years anticipated
  Height is registrated in centimeters and has proven to be of prognostic value in previous research
The primary outcome measure is a prediction model based several factors. One of these is Body Mass Index (BMI). | 2 years anticipated
  BMI is registrated and has proven to be of prognostic value in previous research
The primary outcome measure is a prediction model based several factors. One of these is sports intensity. | 2 years anticipated
  Sports intensity is registrated using the ankle activity score taking type of sports into account and has proven to be of prognostic value in previous research.
The primary outcome measure is a prediction model based several factors. One of these is talar curvature. | 2 years anticipated
  The talar curvature is defined as the angle between the talar neck, most proximal talar part articulating with the tibia and the most distal part of the talus
The primary outcome measure is a prediction model based several factors. One of these is the height of the medial malleolus. | 2 years anticipated
  The medial malleolus is thought to restrict inversion motion, therefore the height is assessed using the angle between the tibiotalar joint and most distal part of the medial malleolus

SECONDARY OUTCOMES:
Inter- and intrarater reliability of the prognostic factors assessed on ankle x-rays | at about 6 months, when 40 patients are included
  Assessment of reliability of the bone geometric factors on anteroposterior and lateral x-rays

OTHER OUTCOMES:
Recurrent ankle sprains and bone geometry | 2 years anticipated
  As all ankle sprains, including recurrent ankle sprains, are recorded, the investigators will perform a subanalysis to assess whether the amount of recurrent ankle sprains is correlated to the bone geometry.
Effect of treatment on development of chronic ankle instability | 2 years anticipated
  Treatment differs per physician and per hospital. Therefore a subanalysis will be performed to assess the influence of treatment on the development of persisting complaints.

CONTACTS AND LOCATIONS:
Locations (4):
- Netherlands (4):
  - Flevoziekenhuis, Almere Stad
  - Slotervaart MC, Amsterdam
  - VUmc, Amsterdam
  - AMC, Amsterdam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pijnenburg AC, Van Dijk CN, Bossuyt PM, Marti RK. Treatment of ruptures of the lateral ankle ligaments: a meta-analysis. J Bone Joint Surg Am. 2000 Jun;82(6):761-73. doi: 10.2106/00004623-200006000-00002. PMID 10859095
- [Background] van Rijn RM, van Os AG, Bernsen RM, Luijsterburg PA, Koes BW, Bierma-Zeinstra SM. What is the clinical course of acute ankle sprains? A systematic literature review. Am J Med. 2008 Apr;121(4):324-331.e6. doi: 10.1016/j.amjmed.2007.11.018. PMID 18374692
- [Background] Milgrom C, Shlamkovitch N, Finestone A, Eldad A, Laor A, Danon YL, Lavie O, Wosk J, Simkin A. Risk factors for lateral ankle sprain: a prospective study among military recruits. Foot Ankle. 1991 Aug;12(1):26-30. doi: 10.1177/107110079101200105. PMID 1959831
- [Background] Mei-Dan O, Kahn G, Zeev A, Rubin A, Constantini N, Even A, Nyska M, Mann G. The medial longitudinal arch as a possible risk factor for ankle sprains: a prospective study in 83 female infantry recruits. Foot Ankle Int. 2005 Feb;26(2):180-3. doi: 10.1177/107110070502600211. PMID 15737262
- [Background] Peduzzi P, Concato J, Kemper E, Holford TR, Feinstein AR. A simulation study of the number of events per variable in logistic regression analysis. J Clin Epidemiol. 1996 Dec;49(12):1373-9. doi: 10.1016/s0895-4356(96)00236-3. PMID 8970487
- [Background] Pavlou M, Ambler G, Seaman SR, Guttmann O, Elliott P, King M, Omar RZ. How to develop a more accurate risk prediction model when there are few events. BMJ. 2015 Aug 11;351:h3868. doi: 10.1136/bmj.h3868. PMID 26264962
- [Background] Ogundimu EO, Altman DG, Collins GS. Adequate sample size for developing prediction models is not simply related to events per variable. J Clin Epidemiol. 2016 Aug;76:175-82. doi: 10.1016/j.jclinepi.2016.02.031. Epub 2016 Mar 8. PMID 26964707
- [Derived] Vuurberg G, Wink LM, Blankevoort L, Haverkamp D, Hemke R, Jens S, Sierevelt IN, Maas M, Kerkhoffs GMMJ. A risk assessment model for chronic ankle instability: indications for early surgical treatment? An observational prospective cohort - study protocol. BMC Musculoskelet Disord. 2018 Jul 18;19(1):225. doi: 10.1186/s12891-018-2124-5. PMID 30021553